CLINICAL TRIAL: NCT00358436
Title: Efficacy and Safety of LAS 34273 in Patients With Moderate to Severe Stable Chronic Obstructive Pulmonary Disease(COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M/34273/31; ACCLAIM II (Other: Almirall,S.A.); CT000742 (Other: Almirall,S.A.)
Record Dates: First submitted 2006-07-28; First posted 2006-07-31 (Estimated); Results first posted 2012-11-01 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Lung function; Exacerbations; Quality of Life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Aclidinium 200 μg once-daily (Experimental): Aclidinium bromide 200 μg once-daily by inhalation
  Interventions: Drug: Aclidinium bromide
- Placebo (Placebo Comparator): Placebo by inhalation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aclidinium bromide — Aclidinium bromide 200 μg once-daily via inhalation by the Eklira Genuair® inhaler: 1 puff in the morning for 52 weeks
  Arms: Aclidinium 200 μg once-daily
Drug: Placebo — Placebo once-daily via inhalation: 1 puff in the morning for 52 weeks
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of LAS 34273 compared to placebo in patients with moderate to severe COPD during one year of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged ≥ 40 years with a clinical diagnosis of moderate to severe stable COPD

Exclusion Criteria:

* History or current diagnosis of asthma, recent respiratory tract infection or acute COPD exacerbation, life expectancy of less than 1 year, known symptomatic prostatic hypertrophy, bladder neck obstruction or narrow-angle glaucoma

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 804 (Actual)
Dates: Start 2006-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, MD, Study Director — AstraZeneca
Locations (120):
- United States (73):
  - Almirall Investigational Sites#926, Jasper, Alabama
  - Almirall Investigational Sites#858, Ozark, Alabama
  - Almirall Investigational Sites#900, Phoenix, Arizona
  - Almirall Investigational Sites#899, Tucson, Arizona
  - Almirall Investigational Sites#855, Tucson, Arizona
  - Almirall Investigational Sites#879, Little Rock, Arkansas
  - Almirall Investigational Sites#932, Carmichael, California
  - Almirall Investigational Sites#904, Encinitas, California
  - Almirall Investigational Sites#903, Fullerton, California
  - Almirall Investigational Sites#930, Los Angeles, California
  - Almirall Investigational Sites#922, Los Angeles, California
  - Almirall Investigational Sites#893, North Hills, California
  - Almirall Investigational Sites#871, Rancho Mirage, California
  - Almirall Investigational Sites#902, Riverside, California
  - Almirall Investigational Sites#850, San Diego, California
  - Almirall Investigational Sites#897, San Diego, California
  - Almirall Investigational Sites#924, Torrance, California
  - Almirall Investigational Sites#882, Walnut Creek, California
  - Almirall Investigational Sites#895, Denver, Colorado
  - Almirall Investigational Sites#880, Fort Collins, Colorado
  - Almirall Investigational Sites#888, Wheat Ridge, Colorado
  - Almirall Investigational Sites#952, Waterbury, Connecticut
  - Almirall Investigational Sites#844, Bay Pines, Florida
  - Almirall Investigational Sites#863, Clearwater, Florida
  - Almirall Investigational Sites#152, DeLand, Florida
  - Almirall Investigational Sites#8533, Melbourne, Florida
  - Almirall Investigational Sites#920, Tamarac, Florida
  - Almirall Investigational Sites#894, Tampa, Florida
  - Almirall Investigational Sites#889, Tampa, Florida
  - Almirall Investigational Sites#890, Atlanta, Georgia
  - Almirall Investigational Sites#907, Decatur, Georgia
  - Almirall Investigational Sites#931, Gainesville, Georgia
  - Almirall Investigational Sites#849, Marietta, Georgia
  - Almirall Investigational Sites#933, Chicago, Illinois
  - Almirall Investigational Sites#872, Hines, Illinois
  - Almirall Investigational Sites#892, River Forest, Illinois
  - Almirall Investigational Sites#864, Evansville, Indiana
  - Almirall Investigational Sites#876, Bowling Green, Kentucky
  - Almirall Investigational Sites#923, Florence, Kentucky
  - Almirall Investigational Sites#866, Lafayette, Louisiana
  - Almirall Investigational Sites#911, Shreveport, Louisiana
  - Almirall Investigational Sites#883, Biddeford, Maine
  - Almirall Investigational Sites#976, Lewiston, Maine
  - Almirall Investigational Sites#843, Baltimore, Maryland
  - Almirall Investigational Sites#868, Cadillac, Michigan
  - Almirall Investigational Sites#884, Minneapolis, Minnesota
  - Almirall Investigational Sites#916, Saint Charles, Missouri
  - Almirall Investigational Sites#906, Butte, Montana
  - Almirall Investigational Sites#909, Omaha, Nebraska
  - Almirall Investigational Sites#846, Cherry Hill, New Jersey
  - Almirall Investigational Sites#885, Newark, New Jersey
  - Almirall Investigational Sites#921, Summit, New Jersey
  - Almirall Investigational Sites#896, Albuquerque, New Mexico
  - Almirall Investigational Sites#861, Chapel Hill, North Carolina
  - Almirall Investigational Sites#919, Charlotte, North Carolina
  - Almirall Investigational Sites#878, Elizabeth City, North Carolina
  - Almirall Investigational Sites#842, Williamston, North Carolina
  - Almirall Investigational Sites#915, Winston-Salem, North Carolina
  - Almirall Investigational Sites#848, Cincinnati, Ohio
  - Almirall Investigational Sites#870, Cincinnati, Ohio
  - Almirall Investigational Sites#847, Columbus, Ohio
  - Almirall Investigational Sites#928, Sylvania, Ohio
  - Almirall Investigational Sites#905, Eugene, Oregon
  - Almirall Investigational Sites#860, Medford, Oregon
  - Almirall Investigational Sites#886, Medford, Oregon
  - Almirall Investigational Sites#910, Charleston, South Carolina
  - Almirall Investigational Sites#918, Greer, South Carolina
  - Almirall Investigational Sites#898, Dallas, Texas
  - Almirall Investigational Sites#854, Fort Worth, Texas
  - Almirall Investigational Sites#875, Houston, Texas
  - Almirall Investigational Sites#881, San Antonio, Texas
  - Almirall Investigational Sites#951, Richmond, Virginia
  - Almirall Investigational Sites#856, Milwaukee, Wisconsin
- Argentina (13):
  - Almirall Investigational Sites#800, Buenos Aires
  - Almirall Investigational Sites#744, Buenos Aires
  - Almirall Investigational Sites#792, Buenos Aires
  - Almirall Investigational Sites#793, Buenos Aires
  - Almirall Investigational Sites#799, Buenos Aires
  - Almirall Investigational Sites#795, Buenos Aires
  - Almirall Investigational Sites#801, Buenos Aires
  - Almirall Investigational Sites#791, Buenos Aires
  - Almirall Investigational Sites#797, El Palomar
  - Almirall Investigational Sites#740, La Plata
  - Almirall Investigational Sites#801, Rosario
  - Almirall Investigational Sites#796, San Miguel de Tucumán
  - Almirall Investigational Sites#794, Vicente López
- Australia (13):
  - Almirall Investigational Sites#807, Adelaide
  - Almirall Investigational Sites#834, Auchenflower
  - Almirall Investigational Sites#808, Bankstown
  - Almirall Investigational Sites#806, Boxhill
  - Almirall Investigational Sites#814, Cairns
  - Almirall Investigational Sites#813, Camperdown
  - Almirall Investigational Sites#811, Carina Heights
  - Almirall Investigational Sites#803, Clayton
  - Almirall Investigational Sites#809, Kippa-Ring
  - Almirall Investigational Sites#8121, Nedlands
  - Almirall Investigational Sites#812, Nedlands
  - Almirall Investigational Sites#805, Toorak Gardens
  - Almirall Investigational Sites#815, Woodville
- Canada (7):
  - Almirall Investigational Sites#823, Edmonton
  - Almirall Investigational Sites#818, Kelowna
  - Almirall Investigational Sites#822, Montreal
  - Almirall Investigational Sites#817, Niagara Falls
  - Almirall Investigational Sites#821, Ottawa
  - Almirall Investigational Sites#935, Ottawa
  - Almirall Investigational Sites#820, Toronto, Ontario
- Mexico (2):
  - Almirall Investigational Sites#827, Monterrey
  - Almirall Investigational Sites#826, Zapopan
- New Zealand (3):
  - Almirall Investigational Sites#936, Auckland
  - Almirall Investigational Sites#830, Grafton
  - Almirall Investigational Sites#832, Tauranga
- South Africa (9):
  - Almirall Investigational Sites#836, Bloemfontain
  - Almirall Investigational Sites#841, Bloemfontein
  - Almirall Investigational Sites#839, Cape Town
  - Almirall Investigational Sites#835, Cape Town
  - Almirall Investigational Sites#837, Cape Town
  - Almirall Investigational Sites#840, Cape Town
  - Almirall Investigational Sites#834, Durban
  - Almirall Investigational Sites#833, eManzimtoti
  - Almirall Investigational Sites#838, Johannesburg

REFERENCES:
- [Derived] Jones PW, Rennard SI, Agusti A, Chanez P, Magnussen H, Fabbri L, Donohue JF, Bateman ED, Gross NJ, Lamarca R, Caracta C, Gil EG. Efficacy and safety of once-daily aclidinium in chronic obstructive pulmonary disease. Respir Res. 2011 Apr 26;12(1):55. doi: 10.1186/1465-9921-12-55. PMID 21518460
- See also: Sponsor web site — http://www.almirall.com/webcorp2/cda/ImD_04_02.jsp
- See also: Co-Sponsor web site — http://www.frx.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in a total of 119 enrolling sites: 72 sites in the United States, 13 sites in Argentina, 13 sites in Australia, 7 sites in Canada, 2 sites in Mexico, 3 sites in New Zealand and 9 sites in South Africa. The first patient was screened in August 2006 and the last patient visit was in June 2008.
Pre-assignment Details: Following a screening visit, patients entered a 14-day run-in period during which they used inhaled salbutamol on an as needed basis. Patients also stopped taking any other COPD medications prohibited by the study protocol. The 14-day run-in period was used to assess the stability of disease and established the patient's baseline characteristics.
Groups:
- Aclidinium Bromide 200 μg Once-daily: Aclidinium bromide 200 μg once-daily by inhalation
Period: Overall Study
Arm/Group | Aclidinium Bromide 200 μg Once-daily | Placebo
Started | 600 | 204
Completed | 446 | 118
Not Completed | 154 | 86
Not completed — Adverse Event | 29 | 13
Not completed — Lack of Efficacy | 34 | 36
Not completed — Lost to Follow-up | 11 | 6
Not completed — Protocol Violation | 8 | 3
Not completed — Withdrawal by Subject | 40 | 17
Not completed — Non-fulfilment of inclusion/exclusion | 4 | 0
Not completed — COPD exacerbation | 22 | 10
Not completed — Other | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aclidinium Bromide 200 μg Once-daily | Placebo | Total
Number analyzed (Participants) | 600 | 204 | 804
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 292 | 85 | 377
  >=65 years | 308 | 119 | 427
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (8.6) | 65.2 (8.6) | 65.2 (8.6)
Gender [Count of Participants; unit: Participants]
  Female | 217 | 80 | 297
  Male | 383 | 124 | 507
Region of Enrollment [Number; unit: participants]
  Argentina | 122 | 42 | 164
  Australia | 70 | 25 | 95
  Canada | 33 | 10 | 43
  Mexico | 7 | 2 | 9
  New Zealand | 12 | 4 | 16
  South Africa | 61 | 20 | 81
  United States | 295 | 101 | 396

OUTCOME MEASURES:

1. Primary Outcome: Trough FEV1 (L) at 28 Weeks on Treatment
Description: Trough FEV1 (mean FEV1 value of the two highest FEV1 readings measured at 23 and 24 hours after inhalation) at 28 weeks
Time Frame: 28 weeks
Population: Intention-to-Treat (ITT) population: all randomised patients who took at least one dose of Investigational Medicinal Product and had at least the baseline and one post-baseline value available for the primary efficacy variable.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Aclidinium Bromide 200 μg Once-daily | Placebo
Number analyzed (Participants) | 594 | 201
Liters | 1.220 (0.008) | 1.162 (0.014)

2. Secondary Outcome: Time to First Moderate or Severe COPD Exacerbation at 52 Weeks on Treatment
Description: Time to first moderate or severe exacerbation: Increase of COPD symptoms during at least 2 consecutive days, treated with antibiotics and/or systemic corticosteroids or an increase in dose of systemic corticosteroids, or leading to hospitalisation.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Aclidinium Bromide 200 μg Once-daily | Placebo
Number analyzed (Participants) | 594 | 201
Days | NA [NA to NA] — The median time to first moderate or severe COPD exacerbation could not be estimated for either group since fewer than 50% of the population had experienced a moderate or severe exacerbation. | NA [NA to NA] — The median time to first moderate or severe COPD exacerbation could not be estimated for either group since fewer than 50% of the population had experienced a moderate or severe exacerbation.

3. Secondary Outcome: Percentage of Patients Who Achieved at Least a 4-unit Decrease From Baseline in the SGRQ Total Score at 52 Weeks on Treatment
Description: Percentage of patients who achieved a clinically relevant improvement in health-related quality of life at 52 weeks, as measured by at least a 4-unit decrease from baseline in St George's Respiratory Questionnaire (SGRQ) total score
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Aclidinium Bromide 200 μg Once-daily | Placebo
Number analyzed (Participants) | 574 | 195
Percentage of Patients
  Yes (% Patients with 4-unit decrease) | 39.0 | 32.8
  No (% Patients without 4-unit decrease) | 61.0 | 67.2

4. Primary Outcome: Trough FEV1 (L) at 12 Weeks on Treatment
Description: Trough FEV1 (mean FEV1 value of the two highest FEV1 readings measured at 23 and 24 hours after inhalation) at 12 weeks
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Placebo: Once daily administered via inhalation
Arm/Group | Aclidinium 200 μg Once-daily | Placebo
Number analyzed (Participants) | 594 | 201
Liters | 1.233 (0.007) | 1.171 (0.012)

ADVERSE EVENTS:
Time Frame: 52 Weeks
Description: Only COPD exacerbations that were fatal or life-threatening are included here. Other COPD exacerbations were not reported as AEs but were included as part of the efficacy evaluations.
Arm/Group | Aclidinium Bromide 200 μg Once-daily | Placebo
Serious Adverse Events (participants affected / at risk) | 62/600 | 23/204
Other Adverse Events (participants affected / at risk) | 445/600 | 136/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aclidinium Bromide 200 μg Once-daily (N=600) | Placebo (N=204)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Acute myocardial infection (Cardiac disorders) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 2 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lobar pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Myocardial infarction (Cardiac disorders) | 5 (5) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 2 (3) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 3 (3) — Two patients, one in each group, reported pneumonia that was considered to be a non-treatment-emergent SAE experienced after discontinuation of study medication.
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) — One patient in the placebo group experienced respiratory failure that was a non-treatment emergent SAE experienced after discontinuation of study medication.
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Haemophilus (Infections and infestations) | 1 (1) | 0 (0)
Rickettsiosis (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple drug overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Open fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulnar fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointerstinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Presycope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Scleroderma renal crisis (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aclidinium Bromide 200 μg Once-daily (N=600) | Placebo (N=204)
Headache (Nervous system disorders) | 85 | 26
Nasopharyngitis (Infections and infestations) | 76 | 23
Upper respiratory tract infection (Infections and infestations) | 65 | 20
Diarrhoea (Gastrointestinal disorders) | 42 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 40 | 15
Urinary tract infection (Infections and infestations) | 29 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 8
Hypertension (Vascular disorders) | 27 | 6
Sinusitis (Infections and infestations) | 27 | 9
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 25 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the information related to this clinical trial is considered strictly confidential and is the property of Almirall. This information will not be given to a third party without the written consent of Almirall. Publication and/or presentation, whether complete or partial, of any part of the data or results of this trial will be subject to revision and written agreement between the investigator and Almirall.